CLINICAL TRIAL: NCT05447273
Title: The Role of Functional Magnetic Resonance Imaging in Preoperative Assessment of Primary Penile Carcinoma
Status: Recruiting | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Marta Daniela Switlyk, Principal Investigator, Oslo University Hospital
Other Study IDs: 428797
Record Dates: First submitted 2022-07-03; First posted 2022-07-07 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Penile Cancer
MeSH Terms: conditions — Penile Neoplasms | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with penile squamous cell carcinoma.: Patients with penile squamous cell carcinoma.
  Interventions: Diagnostic Test: Multi-parametric, functional magnetic resonance imaging (MRI)

INTERVENTIONS:
Diagnostic Test: Multi-parametric, functional magnetic resonance imaging (MRI) — Multi-parametric, functional magnetic resonance imaging (MRI) will be performed in all included patients prior to surgery.

SUMMARY:
The proposed project is intended as a prospective study that includes 60 patients with newly diagnosed penile squamous cell carcinoma (SCC) referred to Oslo University Hospital (OUH), Radiumhospitalet, for surgery, primarily organ-sparing surgery (OSS).

OSS may improve not only quality of life, but also quality of sexual function. However, there is a potential for increased risk of local recurrence after OSS compared to the amputation of the penis. Appropriate preoperative staging, including multi-parametric magnetic resonance imaging (mpMRI), can substantially improve selection of patients and decrease the recurrence rate after surgery.

MpMRI without artificial erection is promising diagnostic tool that is poised to be all-in-one solution for staging and preoperative assessment of primary penile cancer, especially prior to OSS. The method is non-invasive and thus comfortable to perform for most of the patients. Novel MRI techniques are not incorporated into current clinical recommendations, and the potential of new, functional sequences has not been evaluated before. The accuracy of functional, non-erectile mpMRI for detecting and staging of primary penile cancer is not known. Thus, the main purpose of this study is to assess the diagnostic value of this method for preoperative assessment of penile cancer.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed penile squamous cell carcinoma (SCC)
* the patient will benefit from organ-sparing surgery (OSS)
* signed broad consent for cancer research

Exclusion Criteria:

* N/A

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with newly diagnosed penile squamous cell carcinoma (SCC), referred to surgical treatment.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-07-15 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Functional imaging | 2022-2024
  Assess tumor extent and infiltration depth on multi-parametric MRI (mrT-stage) with histopathological evaluation as a reference standard.
  Explore usefulness of multi-parametric MRI in assessing inguinal and pelvic lymph nodes (mrN-stage). 2-fluoro-2-deoxy-D-glucose positron emission tomography/computed tomography (FDG PET-CT), sentinel lymph node evaluation and histopathological examination of the resected specimen will be a gold standard.

SECONDARY OUTCOMES:
Clinical outcome | 2022-2030
  Assess the locoregional recurrence rate and 5-year survival rate following OSS. Clinical outcome data will be obtained from 5 years clinical follow-up at the Department of Urology OUH.
Functional outcome | 2022-2030
  Evaluation of urinary and sexual function following surgery. Functional outcome data will be assessed by urologists using a scoring system and according to the clinical practice, and from interviews with clinical sexologist.

CONTACTS AND LOCATIONS:
Overall Officials: Marta D Switlyk, MD PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hanchanale V, Yeo L, Subedi N, Smith J, Wah T, Harnden P, Bhattarai S, Chilka S, Eardley I. The accuracy of magnetic resonance imaging (MRI) in predicting the invasion of the tunica albuginea and the urethra during the primary staging of penile cancer. BJU Int. 2016 Mar;117(3):439-43. doi: 10.1111/bju.13041. Epub 2015 Jun 3. PMID 25600638
- [Background] Cubilla AL, Barreto J, Caballero C, Ayala G, Riveros M. Pathologic features of epidermoid carcinoma of the penis. A prospective study of 66 cases. Am J Surg Pathol. 1993 Aug;17(8):753-63. doi: 10.1097/00000478-199308000-00001. PMID 8338190
- [Background] Kayes O, Minhas S, Allen C, Hare C, Freeman A, Ralph D. The role of magnetic resonance imaging in the local staging of penile cancer. Eur Urol. 2007 May;51(5):1313-8; discussion 1318-9. doi: 10.1016/j.eururo.2006.11.014. Epub 2006 Nov 13. PMID 17113213
- [Background] Philippou P, Shabbir M, Malone P, Nigam R, Muneer A, Ralph DJ, Minhas S. Conservative surgery for squamous cell carcinoma of the penis: resection margins and long-term oncological control. J Urol. 2012 Sep;188(3):803-8. doi: 10.1016/j.juro.2012.05.012. Epub 2012 Jul 19. PMID 22818137
- [Background] Kieffer JM, Djajadiningrat RS, van Muilekom EA, Graafland NM, Horenblas S, Aaronson NK. Quality of life for patients treated for penile cancer. J Urol. 2014 Oct;192(4):1105-10. doi: 10.1016/j.juro.2014.04.014. Epub 2014 Apr 18. PMID 24747092
- [Background] Romero FR, Romero KR, Mattos MA, Garcia CR, Fernandes Rde C, Perez MD. Sexual function after partial penectomy for penile cancer. Urology. 2005 Dec;66(6):1292-5. doi: 10.1016/j.urology.2005.06.081. PMID 16360459
- [Background] Veeratterapillay R, Teo L, Asterling S, Greene D. Oncologic Outcomes of Penile Cancer Treatment at a UK Supraregional Center. Urology. 2015 May;85(5):1097-1103. doi: 10.1016/j.urology.2014.11.048. Epub 2015 Mar 10. PMID 25769781
- [Background] Petralia G, Villa G, Scardino E, Zoffoli E, Renne G, de Cobelli O, Bellomi M. Local staging of penile cancer using magnetic resonance imaging with pharmacologically induced penile erection. Radiol Med. 2008 Jun;113(4):517-28. doi: 10.1007/s11547-008-0273-6. Epub 2008 May 13. English, Italian. PMID 18478188
- [Background] Scardino E, Villa G, Bonomo G, Matei DV, Verweij F, Rocco B, Varela R, de Cobelli O. Magnetic resonance imaging combined with artificial erection for local staging of penile cancer. Urology. 2004 Jun;63(6):1158-62. doi: 10.1016/j.urology.2004.01.008. PMID 15183971
- [Background] Krishna S, Shanbhogue K, Schieda N, Morbeck F, Hadas B, Kulkarni G, McInnes MD, Baroni RH. Role of MRI in Staging of Penile Cancer. J Magn Reson Imaging. 2020 Jun;51(6):1612-1629. doi: 10.1002/jmri.27060. Epub 2020 Jan 24. PMID 31976600